CLINICAL TRIAL: NCT01566240
Title: A Phase III Multicentre Trial of Weekly Induction Chemotherapy Followed by Standard Chemoradiation Versus Standard Chemoradiation Alone in Patients With Locally Advanced Cervical Cancer
Brief Title: Induction Chemotherapy Plus Chemoradiation as First Line Treatment for Locally Advanced Cervical Cancer
Acronym: INTERLACE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL 11/0034; 2011-001300-35 (EudraCT Number); C37815/A12832 (Other Grant/Funding Number: CRUK)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Chemotherapy; Paclitaxel; Carboplatin; Cisplatin; Radiotherapy; Chemoradiation; Brachytherapy; Stage IB2 Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage IIIB Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Carboplatin; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemoradiation (Active Comparator): Radiotherapy (external beam and brachytherapy) plus concurrent Cisplatin weekly for 5 weeks
  Interventions: Radiation: Radiotherapy; Drug: Cisplatin
- Induction Chemotherapy + Chemoradiation (Experimental): 6 cycles of weekly Paclitaxel and Carboplatin followed by Chemoradiation as per Active Comparator
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 80 mg/m2 (capped at 162mg maximum total dose) weekly for 6 weeks i.e. on days 1, 8, 15, 22, 29 & 36.
  Arms: Induction Chemotherapy + Chemoradiation
Drug: Carboplatin — Carboplatin AUC 2 (capped at 270mg maximum total dose) weekly for 6 weeks i.e. on day 1, 8, 15, 22, 29, & 36.
  Arms: Induction Chemotherapy + Chemoradiation
Radiation: Radiotherapy — Radiotherapy comprising external beam 40-50.4Gy in 20-28 fractions plus intracavity brachytherapy to achieve a minimum total EQD2 dose of 78-86Gy.
Drug: Cisplatin — Cisplatin 40 mg/m2 (capped at 70mg total dose) weekly for five weeks maximum, commencing in the first week of radiotherapy or as soon as blood counts have recovered from induction chemotherapy.

SUMMARY:
Chemoradiation has been the standard treatment for advanced cervical cancer for a decade, but one third of women still die from a failure to control systemic disease. In a recent multicentre phase II trial of 46 women the investigators found that, 68% of women had tumours that responded to weekly induction chemotherapy prior to chemoradiation. The induction chemotherapy had acceptable toxicity and did not compromise the standard chemoradiation treatment. In addition, the overall survival and progression free survival at 3 years was 66% (95% CI 4779). These results, together with acceptable toxicity, provide justification for evaluating induction chemotherapy prior to chemoradiation in a randomised phase III trial. The investigators aim to investigate in a randomised trial whether additional induction chemotherapy given on a weekly schedule immediately before standard chemoradiation leads to an improvement in overall survival. The investigators plan to recruit 770 women with locally advanced cervical cancer who are eligible for standard chemoradiation, they will be randomised to weekly carboplatin and paclitaxel chemotherapy for 6 weeks followed by chemoradiation or to chemoradiation alone. The trial will recruit for 4 years with 5 years of follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed FIGO stage Ib2-IVa squamous, adeno or adenosquamous carcinoma of the cervix (except FIGO IIIA). Patients with histologically confirmed FIGO stage IB1 and positive lymph nodes are also eligible
* Deemed suitable and fit for radical chemoradiation
* Medically fit to receive carboplatin and paclitaxel
* ECOG performance status 0 - 1
* No evidence of active TB
* Aged 18 and over
* Adequate renal function, defined as a GFR ≥ 60 ml/min calculated using the Wright equation (or ≥ 50 ml/min for radioisotope GFR assessment)
* Adequate liver function, as defined by ALT or AST < 2.5 ULN and bilirubin < 1.25 ULN
* Adequate bone marrow function as defined by ANC ≥1.5 x 109/L, platelets ≥ 100 x 109/L
* Using adequate contraception precautions if relevant
* A documented negative HIV test (patients recruited from high risk countries or who have moved within the past 10 years from high risk countries)
* A documented negative pregnancy test (if applicable)
* Capable of providing written or witnessed informed consent

Patients with positive (pelvic/para-aortic/both) nodes (either histologically/PET positive ≥15 mm on CT/MRI) at or below the level of the aortic bifurcation may be included in the study provided none of the exclusion criteria apply.

Exclusion Criteria:

* Previous pelvic malignancy (regardless of interval since diagnosis)
* Previous malignancy not affecting the pelvis (except basal cell carcinoma of the skin) where disease free interval is less than 10 years
* Positive lymph nodes (imaging or histological) above the aortic bifurcation*
* Hydronephrosis which has not undergone ureteric stenting or nephrostomy except where the affected kidney is non-functioning
* Evidence of distant metastasis i.e. any non-nodal metastasis beyond the pelvis
* Previous pelvic radiotherapy
* Prior diagnosis of Crohn's disease or Ulcerative colitis
* Uncontrolled cardiac disease (defined as cardiac function which would preclude hydration during cisplatin administration and any contraindication to paclitaxel)
* Pregnant or lactating * i.e. PET any size, CT/MRI ≥ 15mm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years

SECONDARY OUTCOMES:
Progression free survival | 12 weeks post treatment and then as required
Adverse events (AE) as assessed by the Common Terminology Criteria for Adverse Events v4.03 | To be assessed at every timepoint i.e. baseline; at every chemotherapy cycle, at all follow up visits.
Quality of Life (UK and Ireland only) as assessed by EORTC QLQ-C30, QLQ-CX24 and EQ-5D | Baseline, during induction chemotherapy (Week 4), day 1 of chemoradiation, during chemoradiation (Weeks 3), 4 weeks post end of treatment, and as part of follow up (3 monthly for 2 years; 6 monthly for 3 years until 5 years post randomisation)
Patterns of first relapse (local and/or systemic) | 12 weeks post treatment and as required

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dr McCormack, MBBS, FRCR, Principal Investigator — University College London Hospitals
Locations (35):
- Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil
- India (2):
  - Chittaranjan National Cancer Institute (CNCI), Kolkata
  - Saroj Gupta Cancer Centre and Research Institute, Kolkata
- Istituto Europeo di Oncologia, Milan, Lombardy, Italy
- Instituto Nacional de Cancerologia (INCAN), Mexico City, Mexico
- United Kingdom (30):
  - North Devon District Hospital, Barnstaple, Devon
  - University College London Hospital, London, Greater London
  - Weston Park Hospital, Sheffield, South Yorkshire
  - Belfast City Hospital, Belfast
  - Pilgrim Hospital, Boston
  - Royal Sussex County Hospital, Brighton
  - Velindre Cancer Centre, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Royal Derby Hospital, Derby
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Beatson WOSCC, Glasgow
  - Gloucester Royal Hospital, Gloucester
  - Grantham and District Hospital, Grantham
  - Castle Hill Hospital, Hull
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - St Bart's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - James Cook University Hospital, Middlesbrough
  - Northampton General Hospital, Northampton
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] McCormack M, Eminowicz G, Gallardo D, Diez P, Farrelly L, Kent C, Hudson E, Panades M, Mathew T, Anand A, Persic M, Forrest J, Bhana R, Reed N, Drake A, Adusumalli M, Mukhopadhyay A, King M, Whitmarsh K, McGrane J, Colombo N, Mak C, Mandal R, Chowdhury RR, Alamilla-Garcia G, Chavez-Blanco A, Stobart H, Feeney A, Vaja S, Hacker AM, Hackshaw A, Ledermann JA; INTERLACE investigators. Induction chemotherapy followed by standard chemoradiotherapy versus standard chemoradiotherapy alone in patients with locally advanced cervical cancer (GCIG INTERLACE): an international, multicentre, randomised phase 3 trial. Lancet. 2024 Oct 19;404(10462):1525-1535. doi: 10.1016/S0140-6736(24)01438-7. Epub 2024 Oct 14. PMID 39419054